CLINICAL TRIAL: NCT04339452
Title: Impella-supported Off-pump Coronary Artery Bypass Grafting in High Risk Revascularizations: a Single Center Prospective Observational Study
Brief Title: Impella Supported OPCABG
Status: Active, not recruiting | Type: Observational
Sponsor: Lucian Archambault Durham III (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lucian Archambault Durham III, Lucian Durham, MD, PhD, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Other Study IDs: 37481
Record Dates: First submitted 2020-03-10; First posted 2020-04-09 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Impella 5.5 with SmartAssist Supported OPCABG — Subjects will undergo insertion of an axillary or ascending aortic Impella 5.5 with SmartAssist, followed by Impella-supported OPCABG using a sternotomy approach with shunting of the coronary arteries to achieve myocardial protection.

SUMMARY:
The present study introduces a novel approach to coronary revascularization through the use of a short term minimally-invasive left ventricular assist device (LVAD) to minimize myocardial injury and eliminate low output state during the perioperative period

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Ejection fraction ≤ 35%
* Symptomatic three vessel Coronary Artery Disease with target vessels that are amenable to bypass (as determined by the operating surgeon) or Left main disease
* Adequate Distal target caliber (as determined by the PI or operating surgeon)

Exclusion Criteria:

* Exclusion criteria will include the existing contraindications to either Impella therapy or OPCABG revascularization:

  * Patients with structural heart disease requiring cardiopulmonary bypass
  * Patients with cardiogenic shock who require a period of short-term mechanical circulatory support
  * Patients with mechanical aortic valve
  * Patients with previous median sternotomy
  * Patients with evidence of non-viability on preoperative cardiac MRI or CT scan
  * Insufficient conduit
  * BMI over 50
  * Suspected or known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients fitting inclusion criteria will undergo Impella supported OPCABG using coronary shunts. Inclusion criteria will target patients with ischemic cardiomyopathy, similarly defined to the STICH trial which evaluated coronary revascularization in the setting of heart failure (defined by an EF≤35%). Patients would be considered for enrollment in the setting of symptomatic severe multi-vessel coronary artery disease with target vessels that are amenable to bypass (as determined by the operating surgeon).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hemodynamic stability | Intraoperative
  Intraoperative hemodynamic stability, defined as mean arterial pressure (MAP), cardiac index (CI), central venous pressure (CVP), and cerebral perfusion as measured by NIRS maintained within normal ranges for the entire operative time except potentially for short periods not exceeding 10 minutes in total time.

CONTACTS AND LOCATIONS:
Overall Officials: Lucian A Durham, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No